CLINICAL TRIAL: NCT02711475
Title: "Remove and Discard" Policy in Colonic Diminutive Polyps: is it Always Safe?
Brief Title: Evaluation of Colonic Diminutive Polyps With Electronic Filters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Cardinal Massaia (Other)
Responsible Party: Principal Investigator, carlo verna, M.D., Ospedale Cardinal Massaia
Other Study IDs: OCMAS-1
Record Dates: First submitted 2016-03-08; First posted 2016-03-17 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Diminutive polyps, measuring between 1 and 5 mm, represent the vast majority of colorectal polyps encountered during colonoscopy. Since the chance of harboring advanced adenoma or carcinoma in this kind of polyps is very low, a "remove and discard" technique has been proposed.

The differentiation between adenoma/non adenoma polyps is based on the use of endoscopes equipped with high definition, magnification and optical filters.

DETAILED DESCRIPTION:
Any diminutive polyps encountered during a colonoscopy will be examined with the use of electronic filters and magnification and assigned by the endoscopist to a adenoma/non adenoma category, resected and retrieved: a follow up surveillance period will be assigned on the basis of the endoscopic appearance of the polyps.

Each polyp will then be sent separately to Pathology for the histologic evaluation, and a surveillance interval period will be determined accordingly.

ELIGIBILITY:
Inclusion Criteria:

* All subjects undergoing colonoscopy

Exclusion Criteria:

* Patients assuming oral anticoagulant therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All pationts undergoing screening and non screening colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of accordance between endoscopic and histologic assignment of the polyps to the adenoma/non adenoma category | 1 year
  All the retrieved polyps will be examined and the percentage of accordance between the endoscopic and histologic diagnosis will be determined

SECONDARY OUTCOMES:
Cost savings expressed in dollars between the "remove and discard" technique and histologic examination of samples | 1 year
  The cost of histologic examination for any polyp retrieved will be determined according to the current italian tariff of the procedure and the savings will be calculate
Percentage of concordance between the surveillance periods, determined on the basis of the endoscopic and histologic evaluation of the polyps | 1 year
  For any patient, there will be an analysis of the surveillance period assigned both by the endoscopist and the pathologist in order to determine the percentage of accordance between the two.

CONTACTS AND LOCATIONS:
Overall Officials: CARLO VERNA, M.D., Principal Investigator — CARDINAL MASSAIA HOSPITAL
Locations (1):
- Cardinal Massaia Hospital, Asti, AT, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murino A, Hassan C, Repici A. The diminutive colon polyp: biopsy, snare, leave alone? Curr Opin Gastroenterol. 2016 Jan;32(1):38-43. doi: 10.1097/MOG.0000000000000230. PMID 26574868
- [Background] Repici A, Hassan C, Radaelli F, Occhipinti P, De Angelis C, Romeo F, Paggi S, Saettone S, Cisaro F, Spaander M, Sharma P, Kuipers EJ. Accuracy of narrow-band imaging in predicting colonoscopy surveillance intervals and histology of distal diminutive polyps: results from a multicenter, prospective trial. Gastrointest Endosc. 2013 Jul;78(1):106-14. doi: 10.1016/j.gie.2013.01.035. Epub 2013 Apr 11. PMID 23582472
- [Background] Radaelli F. The Resect-and-Discard Strategy for Management of Small and Diminutive Colonic Polyps. Gastroenterol Hepatol (N Y). 2013 May;9(5):305-8. No abstract available. PMID 23943666
- [Background] Paggi S, Radaelli F, Repici A, Hassan C. Advances in the removal of diminutive colorectal polyps. Expert Rev Gastroenterol Hepatol. 2015 Feb;9(2):237-44. doi: 10.1586/17474124.2014.950955. Epub 2014 Aug 26. PMID 25155348
- [Background] ASGE Technology Committee; Abu Dayyeh BK, Thosani N, Konda V, Wallace MB, Rex DK, Chauhan SS, Hwang JH, Komanduri S, Manfredi M, Maple JT, Murad FM, Siddiqui UD, Banerjee S. ASGE Technology Committee systematic review and meta-analysis assessing the ASGE PIVI thresholds for adopting real-time endoscopic assessment of the histology of diminutive colorectal polyps. Gastrointest Endosc. 2015 Mar;81(3):502.e1-502.e16. doi: 10.1016/j.gie.2014.12.022. Epub 2015 Jan 16. PMID 25597420
- [Result] Rameshshanker R, Wilson A. Electronic Imaging in Colonoscopy: Clinical Applications and Future Prospects. Curr Treat Options Gastroenterol. 2016 Mar;14(1):140-51. doi: 10.1007/s11938-016-0075-1. PMID 26923476